CLINICAL TRIAL: NCT06743009
Title: The Metabolic Effects of the Exercise-metabolite N-lactoyl-phenylalanine (Lac-Phe)
Brief Title: Metabolic Effects of the Exercise-metabolite Lac-Phe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1-10-72-185-23
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-09

CONDITIONS: Healthy Overweight/Obese
Keywords: Lac-Phe; Appetite; Glucose metabolisme
MeSH Terms: conditions — Obesity | interventions — N-lactoyl-phenylalanine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lac-Phe (Experimental): Intravenous infusion of Lac-Phe
  Interventions: Other: N-lactoyl-phenylalanine
- Control (Placebo Comparator): Intravenous infusion of NaCl
  Interventions: Other: NaCl

INTERVENTIONS:
Other: N-lactoyl-phenylalanine — Intravenous infusion of N-lactoyl-phenylalanine (Lac-Phe)
  Other Names: Lac-Phe
  Arms: Lac-Phe
Other: NaCl — 0.9% isotonic NaCl infusion
  Arms: Control

SUMMARY:
The goal of this double-blinded, randomized cross-over clinical trial is to assess the isolated (i.e. outside the context of exercise) effects of Lac-Phe on appetite and glucose concentrations in healthy volunteers with obesity (BMI 28-35).

The main questions it aims to answer are:

* Does Lac-Phe reduce appetite in humans?
* Does Lac-Phe have glucose-lowering properties in humans?

During the study, participants will:

* receive an intravenous infusion of Lac-Phe on one study day and a NaCl infusion on another study day.
* drink a standard mixed meal
* eat an ad libitum meal test
* answer appetite questionnaires
* indirect calorimetry
* blood samples for hormone and substate analyses

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI) between 28-35 kg/m2
* Older than 18 years of age
* Hgb within a normal range (females: 7.3-9.5 mmol/L, males: 8.3-10.5 mmol/L)
* Females can be included if they are either postmenopausal or actively use hormonal contraception (e.g., oral contraceptive pill or hormone-releasing intrauterine device).

Exclusion Criteria:

* Medications affecting glucose metabolism (e.g., Saxenda).
* Anemia
* Diabetes
* Ongoing cancer or other acute/chronic serious diseases (PI will determine)
* Inability to understand Danish or English
* Deemed unsuitable to participate by the PI and co-investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
ad libitum meal test | On the study day, from times 240 minutes and until meal completion as assessed by study participant
  Meal intake (kcal) during the ad libitum meal test

SECONDARY OUTCOMES:
Lac-phe | During the study day, time 0-240 minutes
  plasma concentrations of lac-phe
glucose | During the study day, time 0-240 minutes
  plasma concentrations of glucose
lactate | During the study day, time 0-240 minutes
  plasma concentrations of lactate
c-peptide | During the study day, time 0-240 minutes
  serum concentrations of c-peptide
triglycerider | During the study day, time 0-240 minutes
  plasma concentrations of triglycerides
GLP-1 | During the study day, time 0-240 minutes
  plasma concentration of GLP-1
GIP | During the study day, time 0-240 minutes
  plasma concentrations of GIP
Ghrelin | During the study day, time 0-240 minutes
  plasma concentration of ghrelin
insulin | During the study day, time 0-240 minutes
  serum concentration of insulin
free fatty acids | During the study day, time 0-240 minutes
  Serum concentrations of free fatty acids
LEAP2 | From baseline to end of study day (time 0-240 minutes)
  Plasma concentration of liver-expressed antimicrobial peptide 2 (LEAP2)
Glucagon | From baseline to end of study day (time 0-240 minutes)
  Plasma concentration of glucagon
Gastric emptying assessed by acetaminophen | From baseline to end of study day (time 0-240 minutes)
  Plasma concentration of acetaminophen following oral acetaminophen intake
Subjective appetite - appetite questionaire | Hourly thoughout the study - times 0, 60, 120, 180 and 240 minutes
  We will assess subjective appetite sensations on a visual analog score
Energy expenditure | After 60 and approx 180 minutes
  Indirect calorimetry

CONTACTS AND LOCATIONS:
Locations (1):
- SDCA research laboratory, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
The corresponding author will make data available on reasonable request.